CLINICAL TRIAL: NCT01099709
Title: A Randomized, Open-Label, Single-Center, Single-Dose, Two-Way Crossover Study in Healthy Subjects to Determine the Fed Bioequivalence of Oxycodone Tamper Resistant (OTR) 10-mg Tablets to OxyContin® 10-mg Tablets
Brief Title: A Study to Determine the Fed Bioequivalence of Reformulated OXY Tablets and Original OxyContin® (OXY) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Medical Monitor, Purdue Pharma L.P.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: OTR1002
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-04

CONDITIONS: Healthy Volunteers
Keywords: healthy subjects; opioid
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reformulated OXY 10 mg (Experimental): Reformulated OXY 10 mg x 1 dose
  Interventions: Drug: Reformulated OXY (oxycodone HCl)
- Original OxyContin® (OXY) 10 mg (Active Comparator): Original OxyContin® (OXY) 10 mg x 1 dose
  Interventions: Drug: Original OxyContin® (OXY) (oxycodone HCl)

INTERVENTIONS:
Drug: Reformulated OXY (oxycodone HCl) — Reformulated OXY 10-mg tablet x 1 dose taken with food.
  Arms: Reformulated OXY 10 mg
Drug: Original OxyContin® (OXY) (oxycodone HCl) — Original OxyContin® (OXY) 10-mg tablet x 1 dose taken with food.
  Arms: Original OxyContin® (OXY) 10 mg

SUMMARY:
The purpose of this study is to assess the bioequivalence of a new oxycodone formulation (10 mg) relative to the original OxyContin® (OXY) formulation (10 mg) in the fed state.

DETAILED DESCRIPTION:
Oxycodone hydrochloride (oxycodone) is a semi-synthetic opioid analgesic that is effective in the relief of moderate to severe malignant and non-malignant pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 50, inclusive.
* Body weight ranging from 50 to 100 kg and a BMI ≥18 and ≤34 (kg/m2).
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, and ECG.
* Females of child-bearing potential must be using an adequate and reliable method of contraception.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Any history of or current drug or alcohol abuse for 5 years.
* History of or any current conditions that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of an opioid-containing medication in the past 30 days.
* History of known sensitivity to oxycodone, naltrexone, or related compounds.
* Any history of frequent nausea or emesis regardless of etiology.
* Any history of seizures or head trauma with current sequelae.
* Participation in a clinical drug study during the 30 days preceding the initial dose in this study.
* Any significant illness during the 30 days preceding the initial dose in this study.
* Use of any medication including thyroid hormone replacement therapy (hormonal contraception is allowed), vitamins, herbal, and/or mineral supplements, during the 7 days preceding the initial dose.
* Refusal to abstain from food for 4 hours following administration of the study drugs and to abstain from caffeine or xanthine entirely during each confinement.
* Consumption of alcoholic beverages within 48 hours of initial study drug administration (Day 1) or anytime following initial study drug administration.
* History of smoking or use of nicotine products within 45 days of study drug administration or a positive urine cotinine test.
* Blood or blood products donated within 30 days prior to administration of the study drugs or anytime during the study, except as required by this protocol.
* Positive results for urine drug screen or alcohol screen at Check-in of each period, and HBsAg, HBsAb (unless immunized), anti-HCV.
* Positive Naloxone HCl challenge test.
* Presence of Gilbert's Syndrome or any known hepatobiliary abnormalities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 03-Jan-2007(first study procedure) to 16-Mar-2007(last subject follow-up) at 1 site in the US(Honolulu, HI)
Pre-assignment Details: 145 subjects screened; 48 screen failures; 12 alternates/early discontinuations; 85 randomized; 3 terminated early; 82 completed.
Groups:
- Reformulated OXY (Test): Reformulated OXY 10-mg tablet (test) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations.
- Original OxyContin® (OXY) (Reference): Original OxyContin® (OXY) 10-mg tablet (reference) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations.
Period: Period 1
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Started | 42 | 43
Completed | 41 | 41
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Positive cotinine test | 0 | 1
Not completed — Adverse Event | 1 | 0
Period: Period 2
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Safety Population: Subjects who were randomized, received study drug, and had at least 1 postdose safety assessment.
Arm/Group | Randomized Safety Population
Number analyzed (Participants) | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Bioeqivalence based on Cmax.
Time Frame: Blood samples collected over 72-hour period
Population: Full Analysis Population for PK Metrics. Data from all subjects who were randomized, received study drug, and had at least 1 valid PK metric variable were included in the statistical analysis. Subjects who experienced emesis within 12 hours after dosing were excluded from PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Reformulated OXY (Test): Reformulated OXY 10-mg tablet (test) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion.
- Original OxyContin® (OXY) (Reference): Original OxyContin® (OXY) 10-mg tablet (reference) fed, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion.
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 79 | 81
ng/mL | 14.2 (2.99) | 13.6 (2.75)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — A mixed-model analysis of variance was used to compare (test vs reference) and the 90% confidence intervals were estimated for the ratios (test/reference); Geometric Test/Ref Ratio x 100 = 105, 90% CI 2-sided [101.06 to 108.51] — Bioequivalence was established when 90% Confidence Interval fell within 80%-125%
Statistical Analysis 2: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 105, 90% CI 2-sided [101.06 to 108.51] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

2. Primary Outcome: AUC0-inf - Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over a 72-hour time period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 79 | 81
ng*h/mL | 143 (33.5) | 150 (36.7)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 95.6, 90% CI 2-sided [93.73 to 97.53] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

3. Primary Outcome: AUC0-t - Area Under Plasma Concentration-time Curve From Time Zero to Time of Last Non-zero Plasma Concentration
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72-hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Reformulated OXY (Test): Reformulated OXY 10-mg tablet (test) fed, dosed administered in a two-period, two-sequence, single-dose, two-way crossover fashion.
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 79 | 81
ng*h/mL | 142 (33.4) | 149 (36.6)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric test/Ref Ratio x 100 = 95.7, 90% CI 2-sided [93.85 to 97.68] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

ADVERSE EVENTS:
Time Frame: Ongoing AEs-followed until resolution/30 days after last dose;AEs reported during 7 days following last dose were recorded & followed until resolution,or up to 30 days after last dose. All SAEs were followed until resolution or event/sequelae stabilized.
Description: AEs were learned of through spontaneous reports, subject interview, or subject diaries.
Groups:
- Reformulated OXY 10-mg Tablet (Fed): Reformulated OXY 10-mg tablet (fed) x 1 dose
- Original OxyContin® (OXY) 10-mg Tablet (Fed): Original OxyContin® (OXY) 10-mg tablet (fed) x 1 dose
Arm/Group | Reformulated OXY 10-mg Tablet (Fed) | Original OxyContin® (OXY) 10-mg Tablet (Fed)
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/84
Other Adverse Events (participants affected / at risk) | 41/83 | 29/84
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Reformulated OXY 10-mg Tablet (Fed) (N=83) | Original OxyContin® (OXY) 10-mg Tablet (Fed) (N=84)
Nausea (Gastrointestinal disorders) | 13 (14) | 13/83 (14) — Systematic and nonsystematic assessments were used for reporting AEs.
Dizziness (Nervous system disorders) | 11 (11) | 6 (6) — Systematic and nonsystematic assessments were used for reporting AEs.
Headache (Nervous system disorders) | 9 (11) | 6 (6) — Systematic and nonsystematic assessments were used for reporting AEs.
Somnolence (Nervous system disorders) | 8 (8) | 4 (4) — Systematic and nonsystematic assessments were used for reporting AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days